CLINICAL TRIAL: NCT06390813
Title: Comparison of Square Stepping Exercise Training and Otago Exercise Training in Geriatric Individuals in Terms of Balance and Fear of Falling:Randomized Controlled Studie
Brief Title: Otago Exercises, Square Stepping Exercises, Elderly, Fear of Falling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Huseyin Bilal Ozkadder, Physiotherapist, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10.185.1.79
Record Dates: First submitted 2023-12-29; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Fall; Balance Disorders
Keywords: Square Stepping Exercise; Otago Exercises; Elderly; Fear of Fall; Balance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Square Stepping Exercise (Experimental): It is performed on a thin exercise mat divided into 40 small squares of 250 cm x 100 cm. Individuals are basically required to step in the direction of the length without stepping on the lines forming the squares. Before the CAE training, there will be a 5 minutes warm-up and then a minute cool down period. A total of 18 stepping patterns are planned to be used (6 beginner, 6 intermediate, 6 advanced). Basically, a pattern will be repeated 3-5 times and then the mirror image pattern will be repeated the same number of times. However, if the participant has difficulty in practicing the pattern, it will be repeated until he/she learns it, and after practicing the pattern 3 times without any errors, the next pattern will be used.
  Interventions: Behavioral: Square Stepping Exercise Training
- Otago Exercise Training (Experimental): The exercises were performed 3 days a week for 6 weeks and 18 sessions of 60 minutes in total, including warm-up and cool-down periods of 5 minutes each session. It consists of a total of 22 exercises, including 5 warm-up movements, 5 strengthening exercises and 12 balance exercises.
  Interventions: Behavioral: Otago Exercise Training

INTERVENTIONS:
Behavioral: Otago Exercise Training — A total of 18 sessions of Otago Training were conducted 3 days a week for 6 weeks, each session lasting 60 minutes in total, including 5 minutes of warm-up and cool-down periods.
  Arms: Otago Exercise Training
Behavioral: Square Stepping Exercise Training — A total of 18 sessions of SSE were performed 3 days a week for 6 weeks, each session lasting 40 minutes.
  Arms: Square Stepping Exercise

SUMMARY:
The study was conducted to investigate the effects of Otago Exercise Training and Square Stepping Exercise Training on balance and fear of falling in geriarthric individuals and the superiority of the two exercise training for these parameters. The volunteer individuals participating in the study were randomly divided into 3 groups as otago exercise group, square stepping exercise group and control group with equal number of men and women.

The individuals who participated in study had a homogeneous distribution in terms of age, gender, BMI, height, weight and occupational status in all three groups. However, the number of female individuals was higher in all three groups. In the study, individuals in the exercise training groups received square stepping and otago exercise training 3 days a week for 6 weeks, while individuals in the control group did not receive any training. All three groups were evaluated before and six weeks after the training.

ELIGIBILITY:
Inclusion Criteria:

* 65-75 years old
* Education level at least literate
* Able to walk independently
* Standardized Mini Mental Test Score ≥ 24
* No neurological or lower extremity disease
* Healthy geriatric individuals who agreed to participate in the study

Exclusion Criteria:

* Taking 3 or more medications that may affect cognitive status
* Individuals continuing any exercise/rehabilitation program
* Underwent any surgery for the lower extremities
* Having any neurological-orthopedic problem that may affect gait and balance

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
Tinetti's International Fall Efficacy Scale | 6 weeks
  Asseses perception of balance and stability during activities of daily living. Assesses fear of falling in the elderly population.
  On a scale from 1 to 10, with 1 being very confident and 10 being not confident at all, how confident are you that you do the following activities without falling?
  Score:
  1 = very confident 10 = not confident at all A total score of greater than 70 indicates that the person has a fear of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No